CLINICAL TRIAL: NCT02300207
Title: Electracupuncture Could Ameliorate Orthostatic Intolerance After Weightlessness by Improving Cardiovascular Function
Brief Title: Electroacupuncture is Effective in Cardiac Deconditioning Induced by Head-down Bed Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Jing Sun, Dr., Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LL-2013163
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Cardiovascular Abnormalities; Weightlessness
Keywords: Electroacupuncture; Cardiovascular function; Orthostatic tolerance; Head-down bed rest
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Subjects were in a resting, flat, head-down position -6° from the horizontal. The entire bed rest period was composed of the 4-day head-down bed rest and 2-day period of data collection (before and after the bed rest period). During all of these periods, there was intensive care monitoring. All dining, washing, urination, and defecation were carried out in the bedridden state. Changing position around the body axis was permitted. Dietary intake was 2300-2500 kcal/day, and water intake was 1.0-1.5 L/day. Urine samples (24 h) were collected every day throughout the study. Body weight, heart rate (HR), and blood pressure (BP) were measured in the morning before breakfast.
- Electroacupuncture group (Experimental): During the bed rest phase, subjects in the Electroacupuncture(EA) groups received 30 min of EA treatment, while subjects in the Con group did not receive any treatment.EA was performed using small-sized (1.5 cm) cutaneous electrode pads placed bilaterally at the PC-6 points of the forearms. The intensity of the electrical stimulation was adjusted to produce the most intense tolerable electrical sensation without muscle contractions or uncomfortable feelings at a frequency of 50 Hz using the Hwato electronic acupuncture treatment instrument (Model No. SDZ-II; Suzhou Medical Appliances Co, Ltd, Suzhou, China).
  Interventions: Device: electronic acupuncture treatment instrument

INTERVENTIONS:
Device: electronic acupuncture treatment instrument — Electroacupuncture was performed using small-sized (1.5 cm) cutaneous electrode pads placed bilaterally at the PC-6 points of the forearms (Supplementary Figure 1). The intensity of the electrical stimulation was adjusted to produce the most intense tolerable electrical sensation without muscle contractions or uncomfortable feelings at a frequency of 50 Hz using the Hwato electronic acupuncture treatment instrument (Model No. SDZ-II; Suzhou Medical Appliances Co, Ltd, Suzhou, China).
  Arms: Electroacupuncture group

SUMMARY:
To investigate the changes of cardiovascular function during short-term simulated weightlessness after electroacupuncture (EA) treatment．

DETAILED DESCRIPTION:
Spaceflight is associated with cardiovascular deregulation. However, the influence of microgravity on the cardiovascular system and the underlying mechanisms and countermeasures remain largely unknown. Our previous studies have demonstrated that electroacupuncture (EA) is effective at improving orthostatic tolerance (OT). The purpose of this study was to determine if EA treatment can attenuate cardiovascular deconditioning induced by a 4-day -6° head-down bed rest (HDBR). Fourteen healthy male subjects were randomly allocated into a control group (Con, n=6, 4 days HDBR without countermeasure) and an EA treatment group (EA, n=8, 4 days HDBR with EA at Neiguan [PC-6] for 30 min daily for 4 consecutive days during HDBR). OT was estimated with a combination of +75°/20 min head-up tilt and lower body negative pressure test before and after HDBR. Plasma hormones and heart rate variability were assessed before and after HDBR. Cardiac systolic functions and cerebral blood flow were measured before, during, and after HDBR. The data showed that EA treatment applied daily for 30 min during a 4-day HDBR prevented OT and cardiac systolic function from decrease, prevented autonomic dysfunction (a decrease in the activity of the parasympathetic nervous system), and increased the concentrations of plasma angiotensin II (Ang II) and aldosterone (Ald). These results indicate that 30 min of daily EA treatment at PC-6 is highly effective in partially maintaining OT and cardiac systolic function. Activation of the peripheral sympathetic nervous system and increased plasma hormones is largely responsible for maintaining OT after a 4-day HDBR. Therefore, EA treatment appears to be an effective countermeasure against cardiovascular deconditioning induced by HDBR.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were healthy and physically fit but were not athletes.Comprehensive physical, psychological and routine blood chemistry examinations were performed to select qualified subjects for this research.No medication, smoking, alcohol, or caffeinated drinks were allowed during the study.

Exclusion Criteria:

* skeleton-muscle diseases, visual or acoustic dysfunction, organic and functional diseases of psychiatry and neurology as well as sleep disorders

Ages: 20 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Orthostatic tolerance test | 35 minutes
  The subjects remained at rest in a supine position for 15 min to collect control data, and then tilted to 75° head-up tilt testing (HUT) for 5 second followed by increasing steps of lower body negative pressure (LBNP). LBNP began at -20mm Hg for 5 minutes followed by an increase of -20 mm Hg every 5 minutes until -60 mm Hg (total duration = 20 minutes) or presyncope.

SECONDARY OUTCOMES:
Measurements of cardiac systolic function and cerebral blood flow | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiqing Sun, Ph.D, Study Director — Department of Aerospace Biodynamics, Faculty of Aerospace Medicine, Fourth Military Medical University
Locations (1):
- Department of Aerospace Biodynamics, Faculty of Aerospace Medicine, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Sun J, Li X, Yang C, Wang Y, Shi F, Gao Y, Luan Q, Zhu Y, Sun X. Transcutaneous electrical acupuncture stimulation as a countermeasure against cardiovascular deconditioning during 4 days of head-down bed rest in humans. Acupunct Med. 2015 Oct;33(5):381-7. doi: 10.1136/acupmed-2014-010730. Epub 2015 May 29. PMID 26025383